CLINICAL TRIAL: NCT02730897
Title: Multicentric Analysis of Predictors of N1 Upstaging After Resection of cStage-I NSCLC
Acronym: NUTS
Status: Completed | Type: Observational
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Johnny Moons, Clinical Trial Coordinator, University Hospital, Gasthuisberg
Other Study IDs: NUTS
Record Dates: First submitted 2016-03-21; First posted 2016-04-07 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Surgery; Thoracotomy; VATS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Multicenter Studies as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- VATS: Patients operated by means of minimal invasive technique (VATS or roboticVATS)
  Interventions: Procedure: Central/Peripheral
- Open: Patients operated by means of open thoracotomy
  Interventions: Procedure: Central/Peripheral

INTERVENTIONS:
Procedure: Central/Peripheral — Central versus peripheral location of the primary tumor

SUMMARY:
Five papers showed a lower N1 nodal upstaging with video-assisted thoracic surgery (VATS) compared to open surgery in patients with cStage-I NSCLC . This finding questions the oncologic quality of minimal invasive lung cancer surgery, especially the quality of hilar and intrapulmonary lymh node dissection. However, these retrospective studies did not include analysis of central tumor location, although central tumors have a reported higher chance of N1 upstaging . Possibly, this creates a selection bias as surgeons might select central lesions deliberately for open surgery in line with initial VATS feasibility reports

DETAILED DESCRIPTION:
After optimal preoperative staging, 10 to 25% of patients with clinical stage I (cStage-I) non-small cell lung cancer (NSCLC) are found to have unforeseen positive lymph nodes during resection.

Central tumors, even if they are smaller than 3cm (cT1), have a higher incidence of both intrapulmonary or hilar (N1) or ipsilateral mediastinal (N2) lymph node involvement in comparison to peripheral lesions.

In a cohort of patients that underwent identical preoperative mediastinal evaluation and postoperative pathologic tissue examination of equal quality, nodal upstaging can be used as a quality indicator of oncologic thoracic surgery. Or, it can be used as an instrument to compare different techniques, such as thoracoscopic (VATS) versus open lung resections for lung cancer.

Five papers showed a lower N1 nodal upstaging with video-assisted thoracic surgery (VATS) compared to open surgery. These retrospective studies did not include tumor location.

The investigators hypothesize that this creates a bias as surgeons might have chosen an open approach when the tumor was centrally located. This is in line with initial feasibility reports and guidelines that excluded patients with central lesions. This results in a higher prevalence of positive N1 nodes in patients operated with the open approach.

Our single centre analysis showed a one in three chance of nodal upstaging in central located cStage-I tumors , multivariate analysis showed central location to be the only significant predictor for upstaging, and not the surgical technique.

The aim of this multicentric study is to investigate risk factors for nodal upstaging, including tumor location, in patients with cStage-I NSCLC and validate previous findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated in 2014
* NSCLC on final pathology
* cStage-I (cT1-2a cN0 cM0 ) before start of incision for anatomical resection.
* This includes: open/VATS/ Robotic Assisted Thoracoscopic Surgery (RATS)
* This includes: lobectomy, bilobectomy, sleeve or pneumonectomy (not wedge)

Exclusion Criteria:

* Higher clinical stage than cStage-I
* Former therapy for lung cancer (chemotherapy, radiotherapy, surgery)
* Metastatic disease
* Induction chemo- or radiotherapy
* Non-anatomical resections (wedge)
* Previous lymph node disease
* No positron emission tomography (PET) or Missing PET report

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Per centre, a list of consecutive patients operated for cStage-I NSCLC in 2014 is selected.
  cStage-I is decided based on all information before resection is started in accordance to the 7th edition of TNM
Sampling Method: Non-Probability Sample
Enrollment: 956 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of nodal (N1 and N2) upstaging | immediate postoperative
  Incidence of nodal (N1 and N2) upstaging stratified by 'central' versus 'peripheral' tumor location

SECONDARY OUTCOMES:
Overall Survival | 1 yr postoperative
  To compare survival after resection by open technique or VATS, stratified for the above predictors

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Decaluwé, MD, Study Director — Universitaire Ziekenhuizen KU Leuven

IPD SHARING:
Plan to Share IPD: No